CLINICAL TRIAL: NCT00711659
Title: Standardizing Educational Opportunities on the Complete Pediatric Physical Exam
Acronym: Head to Toe
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Joshua Noe, Assistant Professor, Gastroenterology, Hepatology, and Nutrition, Medical College of Wisconsin
Other Study IDs: PRO00006933
Record Dates: First submitted 2008-07-08; First posted 2008-07-09 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Pediatric Physical Exam
Keywords: Physical exam; Pediatric clerkship; Medical students

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: all third year medical students starting their pediatric clerkship rotation

SUMMARY:
The study proposes that a workshop-based educational experience which utilizes a standardized preceptor training session, a standard skills assessment checklist, and videotaped feedback will improve student comfort and confidence in performing the pediatric physical examination and will provide information to improve the curriculum offerings.

DETAILED DESCRIPTION:
The baseline clinical experience of third year medical students rotating through the clerkship varies, depending on previous clerkships and volunteer opportunities previously encountered. The less experienced third year medical student may require more time and feedback to develop competency. The availability and experience of clinical preceptors and background of the patient may also play a role in the development of pediatric physical examination skills. Other institutions have offered standardized approaches to teaching the health maintenance physical exam. To address these issues, we propose a workshop-based educational experience to (1)determine whether offering a workshop that standardizes exposure to physical exams for junior medical students will improve opportunities to practice physical exam skills in a non-threatening environment, (2)promote immediate feedback to the student that allows for self-reflection by viewing a videotape of their performance, (3)delineate how physical exam skills change in junior medical students throughout the year, and (4)evaluate the inter-rater variability of preceptors teaching health maintenance exams to students rotating through the pediatric clerkship.

ELIGIBILITY:
Inclusion Criteria:

* third year medical students will participate in the physical exam skills workshop as a requirement of their pediatric clerkship; data obtained from review of videotapes of students who consent for data use will be included

Exclusion Criteria:

* data from students who do not consent to use of data will not be used for analysis

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All third year medical students starting their pediatric clerkship at the Medical College of Wisconsin
Sampling Method: Non-Probability Sample
Enrollment: 519 (Actual)
Dates: Start 2007-06; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
To determine if offering a standardized workshop-based education experience for third year medical students will improve student comfort and confidence in performing the pediatric physical exam and provide information to improve curriculum offerings. | 8 weeks (the length of the clerkship rotation)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua D Noe, MD, Principal Investigator — Medical College of Wisconsin; Paola Palma-Sisto, MD, Study Chair — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States